CLINICAL TRIAL: NCT06820606
Title: A Randomized Controlled Trial Comparing Efficacy and Cost Effectiveness of Water Vapour Thermal Therapy (Rezum) and Prostatic Urethral Lift (UroLift) in Men With Benign Prostatic Hyperplasia
Brief Title: Comparing Rezum and Urolift
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHIU Ka Fung Peter, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2024.349-T
Record Dates: First submitted 2025-01-24; First posted 2025-02-11 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rezum (Active Comparator)
  Interventions: Device: Rezum
- UroLift (Active Comparator)
  Interventions: Device: UroLift

INTERVENTIONS:
Device: Rezum — In the REZUM arm, water vapour treatment will be preformed.
  Arms: Rezum
Device: UroLift — In the UroLift arm, prostatic urethral lift treatment will be performed.
  Arms: UroLift

SUMMARY:
This is a randomized controlled trial using a non-inferiority design with the subjects randomized 1:1 to either water vapour thermal treatment (REZUM) arm or prostatic urethral lift (UroLift) arm.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 50 years Symptomatic BPH International prostate symptom score (IPSS) ≥13 Prostate volume 30-80ml

Exclusion Criteria:

* History or high suspicion of prostate cancer
* Current urinary tract infection
* Refractory urinary retention or post-void residual (PVR) ≥250 mL
* Intravesical prostatic protrusion (IPP)>10mm
* Prior prostate surgery
* Known or suspected allergy to nickel, titanium, or polyester/polypropylene
* Urethral stricture, meatal stenosis, bladder neck contracture
* Neurogenic bladder and/or sphincter abnormalities

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in International Prostate Symptom Score (IPSS) at 12 months after treatment | Baseline, 3 months, 6 months and 12 months after intervention
  IPSS score ranging from 0-35 (the higher the worse)

SECONDARY OUTCOMES:
Hospital stays of procedure | From the time patient is hospitalised until the time he discharges
  Measure the hours of in-patient hospitalisation
Number of days on Foley's catheter or self-catheterization after operation | 30 days after intervention
Complication rate | 30 days after intervention
  Assessed by Clavien-Dindo classification
Post-op quality of life score (International Prostate QOL score) | Baseline, 3 months, 6 months and 12 months after intervention
  Change in quality of life assessed by change in International Prostate QOL score (Ranges from 0 to 6; 0 being the best while 6 being the worst)
Post-op quality of life score (EQ5D-5L questionnaire) | Baseline, 3 months, 6 months and 12 months after intervention
  Change in quality of life assessed by Quality of life: EQ5D-5L questionnaire
Change in voiding function in uroflowmetry (Maximum flow rate) | Baseline, 3 months, 6 months and 12 months after intervention
  It is assessed by maximum flow rate (ml/s) in uroflowmetry
Change in voiding function in uroflowmetry (Post void volume) | Baseline, 3 months, 6 months and 12 months after intervention
  It is assessed by post void volume (ml) in uroflowmetry
Post-op erectile function (IIEF-EF) | Baseline, 3 months, 6 months and 12 months after intervention
  Assessed by Erectile function and Ejaculatory function using International Index of Erectile Function Questionnaire - Erectile function domain (IIEF-EF)
Post-op erectile function (MSHQ-EjD-SF) | Baseline, 3 months, 6 months and 12 months after intervention
  Assessed by Erectile function and Ejaculatory function using Male Sexual Health Questionnaire - ejaculatory dysfunction (EjD) Short Form (MSHQ-EjD-SF)
Unplanned readmission rate after operation in 30 days | 30 days after intervention
  Percentage of patients with unplanned readmission
Cost of procedure and related hospitalization | At 12 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ray AF, Powell J, Speakman MJ, Longford NT, DasGupta R, Bryant T, Modi S, Dyer J, Harris M, Carolan-Rees G, Hacking N. Efficacy and safety of prostate artery embolization for benign prostatic hyperplasia: an observational study and propensity-matched comparison with transurethral resection of the prostate (the UK-ROPE study). BJU Int. 2018 Aug;122(2):270-282. doi: 10.1111/bju.14249. Epub 2018 May 6. PMID 29645352
- [Background] Lyauk YK, Jonker DM, Lund TM, Hooker AC, Karlsson MO. Item Response Theory Modeling of the International Prostate Symptom Score in Patients with Lower Urinary Tract Symptoms Associated with Benign Prostatic Hyperplasia. AAPS J. 2020 Aug 27;22(5):115. doi: 10.1208/s12248-020-00500-w. PMID 32856168
- [Background] Elterman D, Shepherd S, Saadat SH, Alshak MN, Bhojani N, Zorn KC, Rijo E, Misrai V, Lajkosz K, Chughtai B. Prostatic urethral lift (UroLift) versus convective water vapor ablation (Rezum) for minimally invasive treatment of BPH: a comparison of improvements and durability in 3-year clinical outcomes. Can J Urol. 2021 Oct;28(5):10824-10833. PMID 34657655
- [Background] Roehrborn CG, Barkin J, Gange SN, Shore ND, Giddens JL, Bolton DM, Cowan BE, Cantwell AL, McVary KT, Te AE, Gholami SS, Moseley WG, Chin PT, Dowling WT, Freedman SJ, Incze PF, Coffield KS, Herron S, Rashid P, Rukstalis DB. Five year results of the prospective randomized controlled prostatic urethral L.I.F.T. study. Can J Urol. 2017 Jun;24(3):8802-8813. PMID 28646935
- [Background] McVary KT, Gange SN, Gittelman MC, Goldberg KA, Patel K, Shore ND, Levin RM, Rousseau M, Beahrs JR, Kaminetsky J, Cowan BE, Cantrill CH, Mynderse LA, Ulchaker JC, Larson TR, Dixon CM, Roehrborn CG. Minimally Invasive Prostate Convective Water Vapor Energy Ablation: A Multicenter, Randomized, Controlled Study for the Treatment of Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia. J Urol. 2016 May;195(5):1529-1538. doi: 10.1016/j.juro.2015.10.181. Epub 2015 Nov 22. PMID 26614889
- [Background] McVary KT, Gittelman MC, Goldberg KA, Patel K, Shore ND, Levin RM, Pliskin M, Beahrs JR, Prall D, Kaminetsky J, Cowan BE, Cantrill CH, Mynderse LA, Ulchaker JC, Tadros NN, Gange SN, Roehrborn CG. Final 5-Year Outcomes of the Multicenter Randomized Sham-Controlled Trial of a Water Vapor Thermal Therapy for Treatment of Moderate to Severe Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia. J Urol. 2021 Sep;206(3):715-724. doi: 10.1097/JU.0000000000001778. Epub 2021 Apr 19. PMID 33872051
- [Background] Teo JS, Lee YM, Ho HSS. An update on transurethral surgery for benign prostatic obstruction. Asian J Urol. 2017 Jul;4(3):195-198. doi: 10.1016/j.ajur.2017.06.006. Epub 2017 Jun 15. PMID 29264231
- [Background] Yip SK, Chan NH, Chiu P, Lee KW, Ng CF. A randomized controlled trial comparing the efficacy of hybrid bipolar transurethral vaporization and resection of the prostate with bipolar transurethral resection of the prostate. J Endourol. 2011 Dec;25(12):1889-94. doi: 10.1089/end.2011.0269. Epub 2011 Sep 16. PMID 21923418
- [Background] Yee CH, Wong JH, Chiu PK, Chan CK, Lee WM, Tsu JH, Teoh JY, Ng CF. Short-stay transurethral prostate surgery: A randomized controlled trial comparing transurethral resection in saline bipolar transurethral vaporization of the prostate with monopolar transurethral resection. Asian J Endosc Surg. 2015 Aug;8(3):316-22. doi: 10.1111/ases.12197. Epub 2015 Jun 3. PMID 26042336
- [Background] Yee CH, Wong JH, Chiu PK, Teoh JY, Chan CK, Chan ES, Hou SM, Ng CF. Secondary hemorrhage after bipolar transurethral resection and vaporization of prostate. Urol Ann. 2016 Oct-Dec;8(4):458-463. doi: 10.4103/0974-7796.192110. PMID 28057992
- [Background] Ng CF, Yee CH, Chan CK, Wong HM, Chiu PK, Tsu JH, Teoh JY, Ho KL. Bipolar transurethral vapourisation versus monopolar transurethral resection of prostate: a randomised controlled trial. Hong Kong Med J. 2017 Jun;23 Suppl 2(3):32-34. No abstract available. PMID 29938669
- [Background] Madersbacher S, Lackner J, Brossner C, Rohlich M, Stancik I, Willinger M, Schatzl G; Prostate Study Group of the Austrian Society of Urology. Reoperation, myocardial infarction and mortality after transurethral and open prostatectomy: a nation-wide, long-term analysis of 23,123 cases. Eur Urol. 2005 Apr;47(4):499-504. doi: 10.1016/j.eururo.2004.12.010. Epub 2005 Jan 23. PMID 15774249
- [Background] Zhang W, Zhang X, Li H, Wu F, Wang H, Zhao M, Hu H, Xu K. Prevalence of lower urinary tract symptoms suggestive of benign prostatic hyperplasia (LUTS/BPH) in China: results from the China Health and Retirement Longitudinal Study. BMJ Open. 2019 Jun 19;9(6):e022792. doi: 10.1136/bmjopen-2018-022792. PMID 31221864